CLINICAL TRIAL: NCT03628495
Title: Effectiveness of a Combined Adequate Pressure and Silicone Intervention in Comparison With Conventional Pressure Therapy for Hypertrophic Scar Treatment: a Randomized Controlled Trial
Brief Title: Effectiveness of a Combined Pressure and Silicone Intervention for Hypertrophic Scar Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSEARS20160418002
Record Dates: First submitted 2018-05-23; First posted 2018-08-14 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Cicatrix, Hypertrophic; Rehabilitation
Keywords: insert; pressure therapy; silicone gel
MeSH Terms: conditions — Cicatrix, Hypertrophic | interventions — Dental Occlusion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The ultrasound data will be processed and the data will be analysed by analysts who are blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SSCP + SPMS (Experimental)
  Interventions: Device: compression; Device: occlusion
- PG (Active Comparator)
  Interventions: Device: compression

INTERVENTIONS:
Device: compression — compression will be delivered using compression garment
Device: occlusion — occlusion will be delivered using silicone gel sheeting
  Arms: SSCP + SPMS

SUMMARY:
Pressure therapy (PT) and silicone therapy are recommended as first-line non-invasive treatments HS, yet the effectiveness of the combination of these two treatments through an RCT trial has not been established yet. This study aims to examine the effectiveness of the combination of adequate pressure therapy and silicone gel sheeting implemented by Smart Scar Care Pad (SSCP) + Smart Pressure Monitored Suit (SPMS) versus conventional Pressure Garment (PG in the management of severe HS in adult. It is hypothesized that the combination of adequate pressure therapy and silicone gel sheeting will demonstrate its superiority in improving scar parameters than conventional pressure garment therapy.

ELIGIBILITY:
Inclusion Criteria:

* The Vancouver Scar Scale (VSS) will be used to screen candidates for the study.10 Isolated scars with a total score of 4 or higher and the score of each item equal to or greater than 1 will be included.
* The scar size should also reach 2*2 cm2 or above to allow adequate area for assessment tool attachement.
* Consenting adult's age between 19 to 60 years old who is able to provide written consent, cooperative, and good compliance with treatment.

Exclusion Criteria:

* the HS area have an open wound or infection;
* the HS have been treated with steroid injections or other intervention (such as traditional Chinese medicine or laser therapy) prior to the study;
* the patients have a medical condition that might affect wound healing (e.g., diabetes mellitus or another serious medical problem);
* the patients with comorbidities that might affect their compliance to treatment: such as severe scar contracture at adjacent area that might be scheduled for reconstructive surgery.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline HS thickness at 6 months | at baseline, one and six month after treatment
  HS thickness measured by the Diagnostic Ultrasound System

SECONDARY OUTCOMES:
Change from baseline HS color at 6 months | at baseline, one and six month after treatment
  HS color measured by the DermaLab Combo Color measurement
Change from baseline HS pliability at 6 months | at baseline, one and six month after treatment
  HS pliability measured by the DermaLab Combo elasticity measurement
Change from baseline HS hydration at 6 months | at baseline, one and six month after treatment
  HS hydration measured by the DermaLab Combo hydration measurement
Itchiness | at baseline, one and six month after treatment
  HS Itchiness measured by the Numerical rating scale
QoL | at baseline, one and six month after treatment
  SF-36 will be used to measure the Quality of Life.

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Li, PhD, Principal Investigator — The Hong Kong Polytechnic University

IPD SHARING:
Plan to Share IPD: No